CLINICAL TRIAL: NCT05955053
Title: The Effect of Childbirth Performed in Collaboration With Midwife-Pregnant Under the Partnership Model on Childbirth Experience and Childbirth Satisfaction: A Randomized Controlled Study
Brief Title: Childbirth Performed in Collaboration With Midwife-Pregnant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Munzur University (Other)
Responsible Party: Principal Investigator, Habibe YAŞAR YETİŞMİŞ, Research assistant, Phd Student, Munzur University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: habibe47
Record Dates: First submitted 2023-06-14; First posted 2023-07-21 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Birth, First; Care Pattern, Maternal; Care; Pregnancy Related
Keywords: Childbirth satisfaction; Midwife-pregnant partnership; Midwife-pregnant cooperation; Childbirth experience; Partnership model; Midwifery; Childbirth; Delivery; Care; Randomized

STUDY DESIGN:
Intervention Model Description: Paralel designed randomized two armed study
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study, in order to minimize the risk of bias, the pregnant women will not know which group they are in, and the statistician will not be informed which group is the intervention and which group is the control during the analysis phase, and the study will be conducted with a blinding method. However, since the person who made the intervention, the researcher (HYY), who took part in the research, is knowledgeable about the intervention and will do the intervention himself, it is not possible to blind the researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midwifery care applied in line with Midwife-Pregnant cooperation (Experimental): The group that received care in line with the midwifery care model checklist
  Interventions: Other: Midwifery care applied in line with Midwife-Pregnant cooperation
- Control group (No Intervention): The group with routine hospital protocol

INTERVENTIONS:
Other: Midwifery care applied in line with Midwife-Pregnant cooperation — Pregnant women who apply to the obstetrics clinic will be informed about the research by the doctor and the pregnant woman whose labor has started will be sent to the delivery room. The researcher will be welcomed by the midwife from the first time the pregnant woman arrives in labor (delivery room), and firstly she will be informed about the purpose of the research and an informative consent form and a pregnant identification form will be filled in that she agrees to participate in the research. During labor and labor, the research midwife (HYY) will be with a pregnant woman until she gives birth and care will be given according to the items in the midwifery care checklist prepared based on the partnership model. After giving birth to a pregnant woman and applying the scales, another pregnant woman will be transferred and care will be given in the same way according to the midwifery care model checklist.
  Arms: Midwifery care applied in line with Midwife-Pregnant cooperation

SUMMARY:
With the medicalization of midwifery care; It has been reported that the autonomy of midwives is reduced, and their relationships with care and care recipients are under threat. For this reason, the midwife had to move away from the concept of being with the woman and face the ideology of being with the institution. In this context, it is thought that there is a need for care models that enable the midwife and woman to work in cooperation. It is thought that establishing a collaborative relationship based on the partnership model between the midwife and the pregnant will be possible with the continuity of care. There are studies in the literature showing that the continuity of midwifery care has positive results at birth. However, no study has been found regarding the partnership or cooperation of the midwife with the pregnant woman during delivery with standards. It is thought that this research to be conducted has a unique value in terms of meeting the need for scientific information on the effect of midwife-pregnant cooperation on birth experience and birth satisfaction. In the study, continuous midwifery care will be given to pregnant women during delivery based on midwife-pregnant cooperation in line with the midwifery care model checklist. It is thought that this midwifery care given during birth will positively affect the birth experience and birth satisfaction.

DETAILED DESCRIPTION:
It has been reported that the medical care model has become widespread, the autonomy of midwives has decreased within the scope of medical care, the care is more medical, the relations of the midwife with the care recipients are under threat and holistic care is avoided. Due to the inability to provide one-to-one holistic care to pregnant women, pregnant women perceive their births as traumatic and experience negative births. In this context, the aim of the research is to evaluate the effect of midwife-pregnant cooperation on birth experience and birth satisfaction within the scope of partnership model. A total of 154 (Intervention; 77, Control; 77) people are planned to be included in the research by performing power analysis. Within the scope of the partnership model, one-to-one care will be given to the pregnant woman in the intervention group during delivery, according to the partnership model, and no intervention will be applied to the control group. Voluntary consent will be obtained from the volunteers to be included in the study and will be randomly included in the groups. Pregnant Information Form, Midwife-Pregnant Collaboration Scale at Birth, Birth Experience Scale, Birth Satisfaction Scale and Midwifery Birth Care Model Checklist will be used to collect research data. Number, percentage distribution, mean and standard deviation, correlation/regression test and t-test for independent groups will be used in the analysis of the research. It is thought that with the care given at the end of the research, the birth experience of the pregnant women will be positive and they will be satisfied with the birth. In the research, it is thought that the positive birth experience and satisfaction of the pregnant women will indirectly give a positive perspective to the normal birth.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35,
* Childbirth started and hospitalized,
* Having a live, single, healthy fetus,
* In the active phase (dilatation= 4 cm and above),
* No maternal and fetal complications that may affect labor,
* At least primary school graduate and no language-communication problem,
* Pregnant women who accepted to participate in the study and whose consent was obtained will be included in the study.

Exclusion Criteria:

* Those with a chronic disease,
* Those with multiparous pregnancy,
* Adolescent pregnant women under the age of 18,
* Advanced age pregnant women over 35 years old,
* Being unable to speak Turkish and having communication difficulties,

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Childbirth Experience | 12 hours after childbirth
  In order to determine the birth experiences of women, the birth experience scale score averages of the pregnant women in the experimental and control groups will be compared. The scale consists of 22 items. The lowest score to be taken from the scale is 22, and the highest score is 88. A high birth experience scale score indicates that the mother had a good birth experience. In this context, at the end of the study, the birth experience scale score averages of both groups will be examined in order to evaluate the birth experience.
Childbirth Satisfaction | 12 hours after childbirth
  In order to determine the birth satisfaction of the women, the mean birth satisfaction scale scores of the pregnant women in the experimental and control groups will be compared. The scale consists of 30 items. The lowest score to be taken from the scale is 30 and the highest score is 150. A high birth satisfaction scale score indicates a high mother's birth satisfaction. In this context, at the end of the study, the mean birth satisfaction scale scores of both groups will be examined in order to evaluate birth satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Munzur University, Tunceli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I can share in case a meta analysis is done

REFERENCES:
- [Background] Boyle S, Thomas H, Brooks F. Women's views on partnership working with midwives during pregnancy and childbirth. Midwifery. 2016 Jan;32:21-9. doi: 10.1016/j.midw.2015.09.001. Epub 2015 Sep 9. PMID 26597110
- [Background] Fleming VE. Women-with-midwives-with-women: a model of interdependence. Midwifery. 1998 Sep;14(3):137-43. doi: 10.1016/s0266-6138(98)90028-6. PMID 9856020
- [Background] Fleming VE. Women and midwives in partnership: a problematic relationship? J Adv Nurs. 1998 Jan;27(1):8-14. doi: 10.1046/j.1365-2648.1998.00474.x. PMID 9515602